CLINICAL TRIAL: NCT03493126
Title: A Pilot Randomized Controlled Trial of Vaginal Estrogen on Postpartum Atrophy, Perineal Pain, and Sexual Function
Brief Title: Vaginal Estrogen on Postpartum Atrophy, Perineal Pain, and Sexual Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: International Urogynecological Association (Other)
Responsible Party: Principal Investigator, Andrew Hundley, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018H0006
Record Dates: First submitted 2018-03-16; First posted 2018-04-10 (Actual); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Vaginal Atrophy
Keywords: postpartum, local estrogen
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estradiol (Experimental): Estrace: pea sized amount 2 times per week from week 1 postpartum to 3 months postpartum.
  Interventions: Drug: Estradiol
- Placebo (Placebo Comparator): Placebo: pea sized amount 2 times per week from week 1 postpartum to 3 months postpartum.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Estradiol — 17β-estradiol vaginal cream
  Other Names: Estrace
  Arms: Estradiol
Other: Placebo — Compounded placebo cream
  Arms: Placebo

SUMMARY:
Pilot randomized, placebo-controlled trial of nulliparous postpartum women with a perineal laceration following a term vaginal delivery comparing vulvovaginal atrophy symptoms between women using vaginal estrogen in the postpartum period with those using placebo.

DETAILED DESCRIPTION:
The overall goal of this study is to determine whether there are benefits to use of low-dose vaginal estrogen in the postpartum period. Dyspareunia and vaginal/perineal pain are well-known sequelae after vaginal delivery. However, the contribution of postpartum vaginal atrophy to these issues is largely unknown. Although the relationship between lactation, relative estrogen deprivation, and vulvovaginal atrophy has been established, there is a paucity of data regarding on the prevalence of vulvovaginal atrophy symptoms in the postpartum period. Additionally, although the benefits of vaginal estrogen in postmenopausal atrophy are well-established, the benefits in the postpartum period are unknown.

ELIGIBILITY:
Inclusion Criteria:

* females >18 years old with at least one prior prenatal care appointment affiliated with The Ohio State University Wexner Medical Center; nulliparous; 1-2 days status post >37 weeks and 0 day vaginal delivery with at least a second degree perineal laceration; English-speaking and able to provide informed consent.

Exclusion Criteria:

* allergies to estradiol cream or its constituents; a vaginal delivery associated with a intrauterine fetal demise or neonatal death; inability to complete questionnaires in English or comply with study protocol; and inability to apply vaginal cream independently. The following medical conditions and diagnoses are also exempted: undiagnosed abnormal vaginal bleeding, known or suspected estrogen-dependent neoplasia, active or history of deep venous thrombosis or pulmonary embolism, active arterial thromboembolic disease, known liver dysfunction or disease, known protein C, protein S, or antithrombin deficiency, or other known thrombophilic disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F Hundley, MD, Principal Investigator — The Ohio State University, Female Pelvic Medicine and Reconstructive Surgery
Locations (1):
- The Ohio State University Urogynecology Clinic, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tennfjord MK, Hilde G, Staer-Jensen J, Ellstrom Engh M, Bo K. Dyspareunia and pelvic floor muscle function before and during pregnancy and after childbirth. Int Urogynecol J. 2014 Sep;25(9):1227-35. doi: 10.1007/s00192-014-2373-2. Epub 2014 Apr 1. PMID 24687365
- [Background] Wisniewski PM, Wilkinson EJ. Postpartum vaginal atrophy. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 2):1249-54. doi: 10.1016/s0002-9378(12)90737-1. PMID 1659199
- [Background] Haran C, van Driel M, Mitchell BL, Brodribb WE. Clinical guidelines for postpartum women and infants in primary care-a systematic review. BMC Pregnancy Childbirth. 2014 Jan 29;14:51. doi: 10.1186/1471-2393-14-51. PMID 24475888
- [Background] Rahn DD, Carberry C, Sanses TV, Mamik MM, Ward RM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen for genitourinary syndrome of menopause: a systematic review. Obstet Gynecol. 2014 Dec;124(6):1147-1156. doi: 10.1097/AOG.0000000000000526. PMID 25415166
- [Background] Eaton AA, Baser RE, Seidel B, Stabile C, Canty JP, Goldfrank DJ, Carter J. Validation of Clinical Tools for Vaginal and Vulvar Symptom Assessment in Cancer Patients and Survivors. J Sex Med. 2017 Jan;14(1):144-151. doi: 10.1016/j.jsxm.2016.11.317. Epub 2016 Dec 20. PMID 28011209

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estradiol | Placebo
Started | 31 | 28
Completed | 28 | 28
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol | Placebo | Total
Number analyzed (Participants) | 31 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (5.1) | 28.0 (4.1) | 28.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: no difference in
  Participants
    Race/Ethnicity: White non-hispanic | 26 | 18 | 44
    Race/Ethnicity: Black non-hispanic | 2 | 3 | 5
    Race/Ethnicity: Hispanic | 1 | 5 | 6
    Race/Ethnicity: Other race/ethnicity | 2 | 1 | 3
    Race/Ethnicity: missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Vulvar Assessment Scale (VUAS)
Description: The VUAS is a four-item measurement administered by a clinical provider that quantifies and rates the patient's responses to questions of dryness, soreness, irritation and pain to external stimulation. Patients are asked whether they have experienced specific symptoms ("yes/no") during the past 4 weeks and rate symptom severity ("none," "mild," "moderate," "severe"). The first 3 items assess dryness, soreness, and irritation during routine activities excluding sexual intercourse and the fourth item assesses pain with external manual stimulation. An option for "no attempt" indicates a patient has not been sexually active within the past 4 weeks. Each item in the VuAS is scored from 0 (none) to 3 (severe) with composite scores calculated by taking the mean of the items when at least two of four items are not missing. Higher scores indicate worse symptoms. The minimum composite score is 0 and maximum composite score is 3.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 31 | 28
score on a scale | 0.10 (0.25) | 0.20 (0.22)

2. Secondary Outcome: Depression
Description: Edinburgh Postnatal Depression Scale (EPDS) The EPDS is a validated 10-question depression assessment for postpartum women, which includes anxiety symptoms and excludes constitutional symptoms associated with depression common in the postpartum period, such as changes in sleeping patterns. Questions 1, 2, & 4 are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3. Questions 3 and 5--10 are reverse scored, with the top box scored as a 3 and the bottom box scored as 0. Minimum total score: 0 Maximum total score: 30. Total score of 10 or higher may be indicative of postpartum depression.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 31 | 28
score on a scale | 4.07 (3.71) | 4.07 (2.99)

3. Secondary Outcome: Urinary Symptoms
Description: Urinary Distress Inventory (UDI-6) The UDI-6 is a questionnaire that includes 6 items evaluating bother from urinary symptoms with higher scores indicating more disability. Each item is scored from 0-3. The total score is the average individual score multiplied by 25. The minimal score is 0 and maximum score is 100.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 31 | 28
score on a scale | 5.6 (10.2) | 10.5 (23.5)

4. Secondary Outcome: Fecal Incontinence
Description: Fecal Incontinence Severity Index (FISI) for bowel symptoms The FISI evaluates patient responses symptom severity to fecal incontinence with higher scores indicating more bothersome anal incontinence symptoms. The FISI score ranges from 0 to 61 with higher score indicating higher severity of the fecal incontinence.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 31 | 28
score on a scale | 16.5 (14.3) | 15.4 (12.4)

5. Secondary Outcome: Sexual Function
Description: Female Sexual Function Index (FSFI) The FSFI is a validated questionnaire to assess sexual function in six domains of sexual function, including desire, arousal, lubrication, orgasm, satisfaction, and pain over the 4 weeks prior to administration of questionnaire with lower scores indicating more sexual dysfunction. The FSFI score ranges from 2-36 with LOWER score indicating worse sexual dysfunction.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 31 | 28
score on a scale | 25.4 (8.1) | 20.5 (10.8)

6. Secondary Outcome: Satisfaction Via Likert Scale
Description: Likert scale Satisfaction will be assessed using the patient satisfaction questionnaire in response to the question, "How satisfied were you with your progress with this treatment?"
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 27 | 27
Participants
  Very satisfied | 14 | 9
  Somewhat satisfied | 5 | 6
  Neutral/unsure | 8 | 11
  somewhat dissatisfied | 0 | 1

7. Secondary Outcome: Adverse Outcomes
Description: At each clinical/research visit the participant will be asked about any adverse events (AEs). AEs will be reported with study outcomes.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 31 | 28
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Estradiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 0/31 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03493126/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03493126/ICF_001.pdf